CLINICAL TRIAL: NCT04496583
Title: Preload Responsiveness as a Signal to Start an Spontaneous Breathing Trial in Mechanically Ventilated Critically Ill Patients
Brief Title: Fluid unLoading On Weaning (FLOW)
Acronym: FLOW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200248
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-01

CONDITIONS: Weaning Failure; Fluid Overload; Cardiac Failure Acute
MeSH Terms: conditions — Edema

STUDY DESIGN:
Intervention Model Description: Randomized prospective controlled study of parallel groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluid Balance Depletive Strategy Group (Active Comparator): Patients with fluid overload under a depletive strategy to attain a predetermined negative balance
  Interventions: Other: Fluid depletion strategy
- Preload Responsiveness Depletive Strategy Group (Experimental): Patients with fluid overload under a depletive strategy to attain a state of preload responsiveness
  Interventions: Other: Fluid depletion strategy

INTERVENTIONS:
Other: Fluid depletion strategy — The fluid depletion strategy will be individualized depending on the response to the standardized furosemide test (one-time dose of 1.0 or 1.5 mg/kg depending on prior furosemide-exposure) with a urinary output (UO) cutoff of 200 ml at 2 hours. The desired depletion endpoint will be targeted by using diuretics (40 mg q6h iv initially, adjusting dose by UO) or ultrafiltration (UF) if UO <200 ml/2h

SUMMARY:
The purpose of this study is to determine if testing preload responsiveness, the normal physiologic state that means that changes in preload determine changes in cardiac output, allows an earlier and physiologically safer weaning from mechanical ventilation in critically ill patients with fluid overload, when compared to a strategy of fluid removal aimed at obtaining a predetermined negative fluid balance.

DETAILED DESCRIPTION:
Fluid overload is a state of global body accumulation of fluids with a deleterious impact in organ function. This condition is frequently found in critically ill patients after acute resuscitation. Its adverse impact is well demonstrated on weaning-induced heart failure, pulmonary and visceral edema, intraabdominal hypertension, etc., which results in longer mechanical ventilation and length of stay, and worse clinical outcomes. Despite these well-known facts, there are no guidelines on how to implement depletive strategies on this phase. The usual approach is to set in advance a desired negative fluid balance for the upcoming days, initiating diuretics or ultrafiltration in preparation for weaning from mechanical ventilation. Unfortunately, this strategy frequently results in excessive and detrimental fluid removal.

A more physiologic approach to guide fluid removal is testing preload responsiveness, which is the normal physiologic state, and means that changes in preload determine changes in cardiac output, with mild or null increment in filling pressures. In contrast, preload unresponsiveness corresponds to a state in which preload increases do not increase stroke volume but produce large increments in filling pressures. This altered state is usually present in patients with fluid overload. Preload responsiveness can be tested routinely in the ICU by assessing the interactions between preload and cardiac output.

Now, in usual clinical practice, weaning from mechanical ventilation is accomplished through a process called the spontaneous breathing trial (SBT), which is a standardized test to mimic the real conditions of breathing without the ventilator, before extubation. One-third of patients fail the initial SBT, which determines a prolonged or difficult weaning and longer stay on mechanical ventilation. Importantly, one of the main determinants of this problem is fluid overload. The pathophysiologic explanation lays in that when switching from positive pressure ventilation to spontaneous breathing, intrathoracic pressure goes from being steadily positive across the ventilatory cycle to markedly negative, promoting increased preload and impeding left ventricular ejection, and this phenomenon is associated to preload unresponsiveness. Interestingly, in most patients with fluid overload, preload responsiveness can be restored just a few hours after starting fluid removal, while modifying fluid balance may take several days. Notably, some patients may persist with preload unresponsiveness even after achieving significant fluid removal.

The investigators hypothesized that in mechanically ventilated patients with fluid overload, a fluid removal strategy aimed at attaining a state of preload responsiveness associates with a decreased incidence of weaning failure from cardiovascular origin, shorter weaning time, and less depletion-induced hypoperfusion events, metabolic derangements and kidney stress compared to patients depleted with a fluid removal strategy aimed at obtaining a predetermined negative fluid balance.

To confirm this hypothesis, the investigators propose a prospective randomized study on 46 critically ill mechanically ventilated patients with fluid overload, comparing these two strategies of depletion and their impact on weaning development and other related systemic functions. Throughout all the protocol, patients will receive general monitoring and management according to ICU standards, plus protocol-specific monitoring that will be added since randomization and before and after SBT attempts, for up to 72 h. Patients will be followed-up for 28 days.

If the investigators' hypothesis is confirmed, it may generate a change in the paradigm of managing fluid overload in critically ill patients, since the physiologic endpoint preload responsiveness may suffice as the valid target and safety parameter to appropriately discontinue mechanical ventilation, shortening the days on mechanical ventilation, the ICU length of stay, and many other costs associated, among additional benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Mechanical ventilation for >24 hours and <7 days
2. Patients who on the daily evaluation to assess their potential for weaning present fluid overload and, in consequence, require fluid depletion before the spontaneous breathing trial
3. Clinical condition resolving or hemodynamically stable condition with acceptable ventilatory status that allows an spontaneous breathing trial according to attending's criteria.

Exclusion Criteria:

1. Pregnancy
2. Do-not-resuscitate status
3. Child B or C liver cirrhosis
4. Circulatory instability
5. Acute coronary syndrome
6. Active bleeding
7. Severe concomitant acute respiratory distress syndrome
8. Malnutrition
9. Muscle weakness severe enough to be considered by itself a risk for weaning failure
10. Patient should be excluded based on the opinion of the clinician/investigator (documented reason)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients on each study group presenting weaning-induced pulmonary edema or weaning failure from cardiovascular origin | 72 hours
  Development of signs of cardiac failure and acute pulmonary edema during the spontaneous breathing trial.
Mean and standard deviation of T time between the starting of fluid depletion and consolidated weaning from mechanical ventilation on each study group. | 7 days
  Time between the starting of fluid depletion and consolidated weaning from mechanical ventilation, measured in hours and days.

SECONDARY OUTCOMES:
Proportion of patients on each study group presenting weaning-induced global and regional hypoperfusion (lactate, capillary refill time, ScvO2, dCO2) | 72 hours
  Development of clinical and laboratory signs of global and regional hypoperfusion due to depletive measures.
Proportion of patients on each study group presenting depletion-induced renal dysfunction assessed by renal stress biomarkers variation. | 72 hours
  Development of laboratory signs of renal compromise due to fluid depletion
Proportion of patients on each study group presenting depletion-induced acid-base and electrolyte disturbances. | 72 hours
  Development of laboratory signs of acid-base and electrolyte derangements due to fluid depletion.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Castro, MD, MPH, Principal Investigator — School of Medicine, Pontificia Universidad Católica de Chile
Locations (1):
- Hospital Clínico UC CHRISTUS, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castro R, Kattan E, Hernandez G, Bakker J. Differential Cardiac Responses after Passive Leg Raising. J Clin Monit Comput. 2024 Oct;38(5):991-996. doi: 10.1007/s10877-024-01180-z. Epub 2024 Jun 6. PMID 38844602